CLINICAL TRIAL: NCT02188823
Title: Examining the Effects of Diet on Health in Prediabetes With an Online Program
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 13-11813p
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Prediabetes
Keywords: prediabetes; obesity; mindful eating; positive affect; low carbohydrate; ketogenic; diet
MeSH Terms: conditions — Prediabetic State; Obesity | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low Carbohydrate Diet (Experimental): Participants will be instructed to follow a low carbohydrate, ketogenic diet: carbohydrate intake 20-35 grams a day not including fiber. Foods permitted include: meats, poultry, fish, eggs, cheese, cream, some nuts and seeds, green leafy vegetables, and most other non-starchy vegetables. Because most individuals self-limit caloric intake, no calorie restriction will be recommended.
  Participants will also be taught information about exercise, sleep, mindfulness, and positive affect practices. The mindfulness-based curriculum will focus on the following elements: training on topics such as mindful meditation, mindful eating, awareness of fullness and hunger signals, and taste satiety. The positive emotion curriculum will include: training on topics such as noticing and savoring positive events, gratitude, positive reappraisal, personal strengths, attainable goals, and acts of kindness.
  Interventions: Behavioral: Low carbohydrate diet

INTERVENTIONS:
Behavioral: Low carbohydrate diet

SUMMARY:
The study is a pilot, designed to provide data regarding the feasibility and acceptability of conducting such a study on a larger scale. The present study is a clinical trial assessing a programs to help people manage prediabetes and lose weight with a low-carbohydrate diet (LC) along with information about positive affect, mindful eating strategies, exercise, and sleep.

DETAILED DESCRIPTION:
Individuals with prediabetes will be assigned to the treatment group. Classes will occur online. Participants will be evaluated at 0, 8, and 16 weeks. Our main outcome of interest is HbA1c (glycated hemoglobin, a measure indicative of blood glucose levels and tied to diabetes severity) at 16 weeks.

ELIGIBILITY:
* Inclusion criteria

  1. Self-reported clinical diagnosis of prediabetes occurring within the past year.
  2. Aged 18 years old and older
  3. Per the Centers for Disease Control and Prevention Diabetes Prevention Recognition Program have a self-reported body mass index (BMI) of ≥ 24 kg/m2 (≥ 22 kg/m2 if Asian).
  4. Willing and able to participate in the intervention such as having sufficient control over their food intake. Must have the ability to make choices about the food they eat; cannot have a lifestyle in which they eat out most of their meals.)
* Exclusion criteria

  1. Unable to provide informed consent.
  2. Non English speaker. The intervention groups are conducted in English.
  3. No current use of insulin, no immediate plans to start or increase diabetic mediations, and no use of diabetes medications besides metformin. Insulin and other diabetes medications other than metformin can alter the safety of the diets, so to ensure greater safety, we will exclude diabetics using insulin or medications besides metformin.
  4. A substance abuse, mental health, or medical condition that, in the opinion of investigators, will make it difficult for the potential participant to participate in the intervention. Such conditions may include: cancer, liver failure, unstable coronary artery disease, severe emphysema, binge eating disorder or history of binge eating disorder, bulimia or strong history of bulimia.
  5. Previous use or recent changes in medications that can interfere with the measures used in the study: current use of insulin; use of systemic (oral or IV) corticosteroids in the 1 month prior to enrollment or severe autoimmune disorders or other conditions (e.g. rheumatoid arthritis, lupus), that are likely to require these medications; and initiation of new class of psychiatric medications in past 2 months. Such medications can alter measures used in our research, such as assessments of markers of inflammation, or negatively influence the safety of the diets.
  6. Pregnant or planning to get pregnant in the next 12 months, breastfeeding or less than 6 months post-partum. The intervention is not designed for the particular diet considerations during pregnancy and breast-feeding.
  7. Current use of weight loss medications or supplements such as Alli or amphetamine-based drugs that are believed to have some effect on weight. Use of weight loss aids by potential participants will be reviewed by a core study team to determine whether participant would be eligible if they stop using the substance.
  8. History of or planned weight loss surgery. The intervention is not designed to address either the often substantial food intake limits that often result from weight loss surgery or the significantly disordered eating that people who fail this extreme intervention may have.
  9. Vegan or vegetarian. The intervention diets are more challenging for vegan and vegetarian participants.
  10. No or very limited internet access at a computer. Must be able to complete the online assessments and access the online class materials.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | baseline to 16 weeks
  We will test whether Hemoglobin A1c changes from pre-intervention to 16 weeks.

SECONDARY OUTCOMES:
Body weight | baseline to 16 weeks
  We will test whether body weight changes from pre-intervention to 16 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- See also: eligibility survey — http://ucbpsych.qualtrics.com/SE/?SID=SV_9LXQ9BJvMR1Qcbb